CLINICAL TRIAL: NCT00851266
Title: A Dose-Escalation, Dose-Ranging Study of the Safety, Tolerability, and Immunogenicity of a Bivalent Influenza Peptide Conjugate Vaccine Formulated With Aluminum- and ISCOMATRIX(TM) Containing Adjuvants (BIPCV/IMX) Evaluated in Healthy Adults 18 to 35 Years of Age
Brief Title: A Study of a Bivalent Influenza Peptide Conjugate Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V512-002; 2009_550
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): V512
  Interventions: Biological: V512
- 2 (Placebo Comparator): Placebo to V512
  Interventions: Biological: Comparator: Placebo to V512

INTERVENTIONS:
Biological: V512 — Subjects received 1 of 8 formulations of the BIPCV/IMX vaccine (V512) in a 3-dose regimen of 0.5 mL injections at Day 1, Month 2, and Month 6:
  1) 0.5 mcg each of A/M2 and B/HA0 peptides with 225 mcg MAA and 20 mcg IMX; 2) 0.5 mcg each of A/M2 and B/HA0 peptides with 225 mcg MAA and 60 mcg IMX; 3) 5 mcg each of A/M2 and B/HA0 peptides with 225 mcg MAA and 20 mcg IMX; 4) 5 mcg each of A/M2 and B/HA0 peptides with 225 mcg MAA and 60 mcg IMX; 5) 5 mcg each of A/M2 and B/HA0 peptides with 225 mcg MAA and 100 mcg IMX; 6) 20 mcg each of A/M2 and B/HA0 peptides with 225 mcg MAA and 20 mcg IMX; 7) 20 mcg each of A/M2 and B/HA0 peptides with 225 mcg MAA and 60 mcg IMX; 8) 20 mcg each of A/M2 and B/HA0 peptides with 225 mcg MAA and 100 mcg IMX;
  Arms: 1
Biological: Comparator: Placebo to V512 — Subjects received placebo to the BIPCV/IMX vaccine (V512) in a 3-dose regimen of 0.5 mL injections at Day 1, Month 2, and Month 6.
  Arms: 2

SUMMARY:
This is a first in man study evaluating the tolerability and immunogenicity of BIPCV/IMX (V512) at increasing concentrations of influenza viral peptides A/M2+B/HA0 peptides and IMX, a saponin-based adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good physical health
* Subject is not in the category of individuals recommended by the CDC to receive influenza vaccine for the upcoming 2 influenza seasons
* Subject agrees not to seek vaccination with licensed influenza vaccines during the study
* Female subjects agree to use acceptable birth control for 6 weeks prior to first dose of vaccine until 1 month post Dose 3

Exclusion Criteria:

* Subject has a history of allergic reaction to the vaccine components
* Subject has has a fever within 3 days of screening
* Subject had a vaccination with an inactive virus within 14 days of Dose 1
* Subject had a vaccination with a live virus within 30 days of Dose 1

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety: Safety and tolerability of BIPCV/IMX as assessed by vaccine-related SAEs; Immunogenicity: 1) A/M2 specific immunogenicity; 2) B/HA0 specific immunogenicity | Safety: 7 months; Immunogenicity: 1) 7 months; 2) 7 months

SECONDARY OUTCOMES:
Persistence of A/M2 and B/HA0 immunogenicity | Months 12, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC